CLINICAL TRIAL: NCT06576362
Title: Anatomopathological Evaluation of a New Ultrasound-guided Transuterine Vaginal Biopsy Technique in Uterine Fibromatous Disease
Brief Title: Evaluation of Ultrasound-guided Transuterine Vaginal Biopsy Technique in Uterine Fibromatous Disease
Acronym: EFIBIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM23-0387; 2024-A01337-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Fibroid; Uterine Corpus Smooth Muscle Neoplasm
Keywords: TMM; BVTE; diagnosis; Vaginal biopsy; echo-guided transuterine vaginal biopsy; myomectomy; hysterectomy
MeSH Terms: conditions — Leiomyoma; Disease | interventions — Hysterectomy

STUDY DESIGN:
Intervention Model Description: Prospective diagnostic study vs. reference technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Echoguided transuterine vaginal biopsy (Experimental): Echoguided transuterine vaginal biopsy on women presenting to hospital with a surgical indication for myomectomy or hysterectomy
  Interventions: Procedure: Echoguided transuterine vaginal biopsy performed before myomectomy or hysterectomy

INTERVENTIONS:
Procedure: Echoguided transuterine vaginal biopsy performed before myomectomy or hysterectomy — Echoguided transuterine vaginal biopsy performed before myomectomy or hysterectomy

SUMMARY:
The goal of this diagnostic, prospective study is to evaluate an innovative, minimally invasive surgical technique for diagnosing uterine smooth muscle tumors by biopsy, in women aged 18 and more, and to evaluate complications relating to the the technique and its potential adverse events.

Participants presenting at hospital patients presenting a surgical indication for myomectomy or hysterectomy during the inclusion period will be offered the study.

Preoperatively, women will undergo the following two examinations:

1. A pelvic MRI, the characteristics of which will be analyzed by the expert women's imaging team.
2. A BVTE under general anaesthetic in the operating theatre on the day of the planned myomectomy or hysterectomy.

250 women will be included in this study within a periofd of inclusion of 36 months and their participation is estimated to 7 months Total study duration is 43 months

DETAILED DESCRIPTION:
Fibroma is the most common uterine smooth muscle tumor. Women are symptomatic in 30% of cases. A large proportion of fibroids are asymptomatic and discovered on imaging. Surgical management is the only recommended first-line treatment option in cases of symptoms. Hysterectomy is the most radical treatment, but for women wishing to preserve their fertility, myomectomy is the most suitable option. This is performed by hysteroscopy, laparoscopy or laparotomy. The main risk of myomectomy is massive intraoperative haemorrhage, requiring blood transfusion or even a haemostasis hysterectomy. There are non-surgical alternatives using embolization and radiofrequency, but these techniques do not provide a definitive diagnosis of fibroids, as they do not involve histological sampling.

The benign uterine fibroma is part of the broader concept of uterine smooth muscle tumors, which also includes myometrial malignancies of varying malignancy (uterine sarcomas, cellular fibromas, STUMP (Uterine smooth muscle tumors of uncertain malignant potential)).

Magnetic resonance imaging (MRI) is the most effective examination for discriminating fibroids from TMM, but its reliability is limited. This leads to inappropriate management in a number of situations. The first is the risk of over-treatment by performing surgery for suspected TMM on MRI in a patient with few or no symptoms and a final histological diagnosis of fibroid. The second is the risk of unsatisfactory, even deleterious, carcinological surgical treatment in a symptomatic patient with a reassuring MRI diagnosis but a final histological diagnosis of TMM. The last situation is the possibility of treating a lesion labelled fibroid on MRI with an alternative technique (embolization, radiofrequency, HIFU) when it is in fact a TMM, thereby delaying appropriate management and worsening the prognosis.

Ultrasound-guided transuterine vaginal biopsy (ETVB) is an innovative and promising minimally invasive technique for preoperative anatomopathological diagnosis. It can be used to obtain a histological diagnosis, thus avoiding the need for surgery and the inappropriate treatment described above Primary objective: To validate an innovative, minimally invasive surgical technique for diagnosing uterine smooth muscle tumors by biopsy.

Secondary objectives Evaluate the complications associated with the technique, as well as its potential adverse effects.

Exploratory objectives: To assess the feasibility of the technique in routine practice.

Primary endpoint: Estimation of the anatomopathological sensitivity of BVTE, with its 95% confidence interval, by comparing it with the reference technique, i.e. anatomopathological diagnosis on surgical specimen, to ensure a low number of false negatives (fibroid diagnosis on BVTE with final diagnosis of TMM).

Secondary endpoints: Estimation of specificity, positive and negative predictive values and likelihood ratios of BVTE, with their confidence intervals, number of intraoperative and postoperative complications according to the Clavien-Dindo classification.

Exploratory criteria if applicable: Evaluation of equipment availability, cost, simplicity of performance as assessed by the operator.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age consulting at the hospital who require surgical management for uterine smooth muscle tumors (fibroma or TMM).
2. Able to give written consent
3. Beneficiary or beneficiary of a social security scheme

Exclusion Criteria:

1. Person in a period of exclusion from another research protocol at the time consent is signed.
2. Subjects covered by articles L1121-5 to 1121-8 of the French Public Health Code, i.e. :

   * Pregnant women, parturients and nursing mothers
   * Persons deprived of their liberty by judicial or administrative decision
   * Persons subject to psychiatric monitoring under articles L3112-1 and L3113-1 who are not covered by the provisions of article L1121-8.
   * Minors
   * Adults subject to a legal protection measure or unable to express their consent.
3. A person who does not have a sufficient command of the French language to be able to give consent to participate in research.
4. Any other reason which, in the opinion of the investigator, could compromise the safety of the research participant and/or interfere with the evaluation of the research objectives.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women over 18 years of age consulting at the hospital, who require surgical management for uterine smooth muscle tumors (fibroma or TMM).
Enrollment: 250 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Validate an innovative, minimally invasive surgical technique for diagnosing uterine smooth muscle tumors by biopsy | From enrollment before surgery to the follow-up visit 3 months after surgery
  Estimate the anatomopathological sensitivity of BVTE, with its 95% confidence interval, by comparing it with the reference technique, i.e. anatomopathological diagnosis on surgical specimens, to ensure a low number of false negatives (fibroid diagnosis on BVTE with final diagnosis of TMM)

CONTACTS AND LOCATIONS:
Overall Officials: Laura MIQUEL, Dr, Principal Investigator — Assistance Publique - Hôpitaux de marseille

IPD SHARING:
Plan to Share IPD: No